CLINICAL TRIAL: NCT06129162
Title: A Comparison of Pain Perception for Nerve Block and Infiltration Injection Using the Conventional Method and Two Computerized Control Systems
Brief Title: Pain Perception Comparison of Computerized vs Conventional Injection Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Osamah Mohammed Abdulghani Almekhlafi, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A0108023PP
Record Dates: First submitted 2023-10-20; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Pain Perception; Local Anesthesia
Keywords: Pain perception; Inferior Alveolar Nerve; Infiltration; Local Anesthesia; STA Single Tooth Anesthesia® System; Star Pen anesthesia device; Conventional syringe

STUDY DESIGN:
Intervention Model Description: Selected children will be divided randomly into 3 groups:
  * Control group (Group I).
  * STA group (Group II).
  * Star pen group (Group III).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: Control Group (Active Comparator): Use a conventional syringe to inject anesthetic solution by the inferior alveolar nerve block (IANB) technique. Also, use a conventional syringe to inject anesthetic solution by buccal infiltration (BI) technique.
  Interventions: Device: STA Single Tooth Anesthesia® System.; Device: Star Pen anesthesia device.
- Group II: STA group (Experimental): Use STA Wand® (CCLA) to inject anesthetic solution by the inferior alveolar nerve block (IANB) technique. Also, use STA Wand® (CCLA) to inject anesthetic solution by buccal infiltration (BI) technique.
  Interventions: Device: Conventional Syringe; Device: Star Pen anesthesia device.
- Group III: Star pen group (Experimental): Use a Star Pen device to inject anesthetic solution by the inferior alveolar nerve block (IANB) technique. Also, use a Star Pen device to inject anesthetic solution by buccal infiltration (BI) technique.
  Interventions: Device: Conventional Syringe; Device: STA Single Tooth Anesthesia® System.

INTERVENTIONS:
Device: Conventional Syringe — Dental local anesthesia injection is given by conventional syringe by two injection methods inferior alveolar nerve block and buccal infiltration.
  Arms: Group II: STA group; Group III: Star pen group
Device: STA Single Tooth Anesthesia® System. — Dental local anesthesia injection is given by STA device by two injection methods inferior alveolar nerve block and buccal infiltration.
  Arms: Group I: Control Group; Group III: Star pen group
Device: Star Pen anesthesia device. — Dental local anesthesia injection is given by Star Pen anesthesia device by two injection methods inferior alveolar nerve block and buccal infiltration.
  Arms: Group I: Control Group; Group II: STA group

SUMMARY:
This study was conducted to a Comparison of Pain Perception for Nerve Block and Infiltration Injection Using the Conventional Method and Two Computerized Control Systems.

DETAILED DESCRIPTION:
The study evaluates and compares pain perception of the inferior alveolar nerve block (IANB) and buccal infiltration anaesthetic in children using a Conventional syringe, STA Single Tooth Anesthesia® System and Star Pen anaesthesia device.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy children (5-8) years old, and free from systemic diseases.
2. Children who require local anesthetic injection for any dental treatment.
3. Cooperative children (positive or definitely positive on Frankel's scale).
4. Children who have no contraindications to the usage of selected local anesthetic agents.

Exclusion Criteria:

* All that does not correspond to inclusion criteria.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
scale of pain perception by Wong-Baker FACES Pain Rating scale | Up to 12 weeks.
  The primary outcome was evaluated using Wong-Baker FACES Pain Rating scale. The child was briefly explained about each face and then asked to select the face that best described their feelings during the administration of local anesthesia. The scale consists of 6 cartoon faces depicting varying facial expressions, ranging from a very happy face (score 0) to a very sad one (score 10).
scale of pain perception by Sounds, eyes, and motor (SEM) scale. | Up to 12 weeks.
  The primary outcome was evaluated using Sounds, eyes, and motor (SEM) scale. These responses are categorized on a scale ranging from 1-4 categories comfort, mild discomfort, moderately painful, and painful. Two pediatric dentists who are blind to injection devises will conduct the clinical evaluation. A third examiner will be consulted if there is a disagreement between the results of the first two.

CONTACTS AND LOCATIONS:
Overall Officials: Osamah M Almekhlafi, Master, Principal Investigator — Researcher of Pediatric Dentistry Faculty of Dentistry Mansoura University; Salwa M Awad, Prof, Study Director — Prof. of Pediatric Dentistry and Dental Public Health Faculty of Dentistry Mansoura University; Rizk A Elagamy, PhD, Study Director — Assistant Professor of Pediatric Dentistry Faculty of Dentistry Mansoura University
Locations (1):
- Faculty of dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol to other researchers
Supporting Information: Study Protocol
Time Frame: within 6 month
Access Criteria: for anyone